CLINICAL TRIAL: NCT02605291
Title: The Effect of Dietary Macronutrient Manipulation and Glycogen Depleting Exercise on Substrate Oxidation at Rest and During Exercise
Brief Title: Dietary Macronutrient Manipulation and Substrate Oxidation During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Lucozade Ribena Suntory (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ERN_15-0963
Record Dates: First submitted 2015-11-06; First posted 2015-11-16 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Dietary Manipulation
MeSH Terms: interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental arm 1 (Experimental): One of three 7-day study arms consisting of 3 days of standardised diet followed by 3 days of dietary macronutrient manipulation and 1 day of experimental testing.
  Interventions: Other: Diet with a different macronutrient content A; Other: Interval treadmill running exercise; Other: Steady state treadmill running exercise
- Experimental arm 2 (Experimental): One of three 7-day study arms consisting of 3 days of standardised diet followed by 3 days of dietary macronutrient manipulation and 1 day of experimental testing.
  Interventions: Other: Diet with a different macronutrient content B; Other: Interval treadmill running exercise; Other: Steady state treadmill running exercise
- Experimental arm 3 (Experimental): One of three 7-day study arms consisting of 3 days of standardised diet followed by 3 days of dietary macronutrient manipulation and 1 day of experimental testing.
  Interventions: Other: Diet with a different macronutrient content C; Other: Interval treadmill running exercise; Other: Steady state treadmill running exercise

INTERVENTIONS:
Other: Diet with a different macronutrient content A — A diet with altered macronutrient content will be provided to participants on days 4-6 of experimental arm 1.
  Arms: Experimental arm 1
Other: Diet with a different macronutrient content B — A diet with a different macronutrient content compared to arm 1 will be provided to participants on days 4-6 of experimental arm 2.
  Arms: Experimental arm 2
Other: Diet with a different macronutrient content C — A diet with a different macronutrient content compared to arms 1 and 2 will be provided to participants on days 4-6 of experimental arm 3.
  Arms: Experimental arm 3
Other: Interval treadmill running exercise — Participants will perform interval treadmill running exercise on days 4 and 5 of all experimental arms.
Other: Steady state treadmill running exercise — Participants will perform steady state treadmill running exercise on day 7 of all experimental arms.

SUMMARY:
This study will investigate the effect of dietary macronutrient manipulation on glycogen (stored carbohydrate) levels in the muscle and substrate oxidation during exercise. The investigators will investigate the hypothesis that manipulating the macronutrient content of the diet will alter the levels of glycogen in the muscle and, in turn, substrate oxidation during exercise.

DETAILED DESCRIPTION:
One way to help reduce body fat is to expend more energy from the oxidation of fat as a fuel. Exercise is one way to increase fat oxidation. The extent to which exercise facilitates the use of fat as a fuel may be influenced by an individual's dietary intake.

This study aims to establish the effect of dietary macronutrient manipulation on muscle glycogen levels and substrate oxidation during exercise. Participants will undertake three separate trial periods. During each trial period participants will consume a diet containing different macronutrient compositions. For each of the trials the investigators will assess how the macronutrient composition of the diet affects muscle glycogen level and substrate oxidation during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Non-smoking - currently and for the past 5 years
* Fitness - V̇O2max 40-60 ml/kg/min
* Body mass index (20-25 kg/m2)

Exclusion Criteria:

* Known or suspected intolerance to the dietary interventions or their stated ingredients.
* Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.
* Previous participation in this study.
* Recent history (within the last year) of alcohol or other substance abuse.
* An employee of the sponsor or the study site or members of their immediate family.
* Abnormal / extreme habitual dietary practice / intake
* Recent (≤3 months) dietary practice that may be deemed as low and/or high in macronutrients will be excluded.
* The taking of any prescribed medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Muscle glycogen concentration after dietary macronutrient manipulation | Day 7 of all experimental arms
  Muscle glycogen concentration will be measured after the dietary macronutrient manipulation intervention.

SECONDARY OUTCOMES:
Rate of fat oxidation at rest (g/min) | For 20 min on Day 7 of all experimental arms
  Whole body oxygen consumption (VO2, L/min) and carbon dioxide production (VCO2, L/min) at rest will be measured using indirect calorimetry to calculate the rate of fat oxidation at rest (g/min).
Rate of fat oxidation during exercise (g/min) | During 60 min of exercise on day 7 of all experimental arms
  Whole body oxygen consumption (VO2, L/min) and carbon dioxide production (VCO2, L/min) during exercise will be measured using indirect calorimetry to calculate the rate of fat oxidation during exercise (g/min).
Rate of carbohydrate oxidation at rest (g/min) | For 20 min on Day 7 of all experimental arms
  Whole body oxygen consumption (VO2, L/min) and carbon dioxide production (VCO2, L/min) at rest will be measured using indirect calorimetry to calculate the rate of carbohydrate oxidation at rest (g/min).
Rate of carbohydrate oxidation during exercise (g/min) | During 60 min of exercise on day 7 of all experimental arms
  Whole body oxygen consumption (VO2, L/min) and carbon dioxide production (VCO2, L/min) during exercise will be measured using indirect calorimetry to calculate the rate of carbohydrate oxidation during exercise (g/min).
Blood glucose concentration | At 0, 20, 40 and 60min into exercise on day 7 of all experimental arms.
  Blood glucose concentration will be assessed in blood samples taken during exercise.
Blood insulin concentration | At 0, 20, 40 and 60min into exercise on day 7 of all experimental arms
  Blood insulin concentration will be assessed in blood samples taken during exercise.
Blood fatty acid concentration | At 0, 20, 40 and 60min into exercise on day 7 of all experimental arms
  Blood fatty acid concentration will be assessed in blood samples taken during exercise.
Change in intramuscular triglyceride (IMTG) content after exercise | IMTG content measured just before and immediately after 60min of exercise on Day 7 of all experimental arms
  IMTG utilisation during exercise (or change in IMTG content pre-post exercise) will be measured by comparing the IMTG content before and after exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Gareth A Wallis, PhD, Principal Investigator — University of Birmingham
Locations (1):
- School of Sport Exercise and Rehabilitation Sciences, University of Birmingham, Birmingham, United Kingdom